CLINICAL TRIAL: NCT04620330
Title: A Phase 2 Study of Avutometinib (VS-6766) (Dual RAF/MEK Inhibitor) as a Single Agent and In Combination With Defactinib (FAK Inhibitor) in Recurrent KRAS-Mutant (KRAS-MT) and BRAF-Mutant (BRAF-MT) Non-Small Cell Lung Cancer (NSCLC) (RAMP 202)
Brief Title: A Study of Avutometinib (VS-6766) + Defactinib in Recurrent KRAS G12V, Other KRAS and BRAF Non-Small Cell Lung Cancer
Acronym: RAMP202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-202
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer; KRAS Activating Mutation
Keywords: NSCLC; KRAS-G12V; G12V; BRAF; V600E; KRAS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: avutometinib (VS-6766) monotherapy (Experimental): in patients with NSCLC KRAS-G12V tumor
  Interventions: Drug: avutometinib (VS-6766)
- Arm 2: avutometinib (VS-6766) in combination with defactinib (Experimental): in patients with a NSCLC KRAS-G12V tumor
  Interventions: Drug: avutometinib (VS-6766) and Defactinib
- Arm 3: avutometinib (VS-6766) in combination with defactinib (Experimental): in patients with a NSCLC KRAS-other (non-G12V) tumor
  Interventions: Drug: avutometinib (VS-6766) and Defactinib
- Arm 4: avutometinib (VS-6766) in combination with defactinib (Experimental): in patients with a NSCLC BRAF-V600E tumor
  Interventions: Drug: avutometinib (VS-6766) and Defactinib
- Arm 5:avutometinib (VS-6766) in combination with defactinib (Experimental): in patients with a NSCLC BRAF-non-V600E tumor
  Interventions: Drug: avutometinib (VS-6766) and Defactinib

INTERVENTIONS:
Drug: avutometinib (VS-6766) — Monotherapy
  Arms: Arm 1: avutometinib (VS-6766) monotherapy
Drug: avutometinib (VS-6766) and Defactinib — Combination therapy
  Other Names: avutometinib (VS-6766) and VS-6063
  Arms: Arm 2: avutometinib (VS-6766) in combination with defactinib; Arm 3: avutometinib (VS-6766) in combination with defactinib; Arm 4: avutometinib (VS-6766) in combination with defactinib; Arm 5:avutometinib (VS-6766) in combination with defactinib

SUMMARY:
This study will assess the safety and efficacy of avutometinib (VS-6766) monotherapy or VS-6766 in combination with defactinib in subjects with recurrent Non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 2 study designed to evaluate safety and tolerability and efficacy of avutometinib (VS-6766) versus avutometinib (VS-6766) in combination with defactinib in subjects with KRAS and BRAF mutant NSCLC following treatment with an appropriate platinum-based regimen and an approved immune checkpoint inhibitor (CPI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age
* Histologic or cytologic evidence of NSCLC
* Known KRAS or BRAF mutation
* The subject must have received appropriate prior therapy
* Measurable disease according to RECIST 1.1
* An Eastern Cooperative Group (ECOG) performance status ≤ 1
* Adequate organ function
* Adequate recovery from toxicities related to prior treatments
* Agreement to use highly effective method of contraceptive

Exclusion Criteria:

* Systemic anti-cancer therapy within 4 weeks of the first dose of study therapy
* History of prior malignancy, with the exception of curatively treated malignancies
* Major surgery within 4 weeks (excluding placement of vascular access)
* History of treatment with a direct and specific inhibitor of MEK, KRAS or BRAF except for treatment of BRAF V-600E mutant NSCLC
* Exposure to strong CYP2C9 and CYP3A4 inhibitors or inducers within 7 days prior to the first dose and during the course of therapy
* Symptomatic brain metastases requiring steroids or other local interventions.
* Known SARS-Cov2 infection ≤28 days prior to first dose of study therapy
* Active skin disorder that has required systemic therapy within the past 1 year
* History of rhabdomyolysis
* Concurrent ocular disorders
* Concurrent heart disease or severe obstructive pulmonary disease
* Subjects with the inability to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
To determine the optimal regimen, either avutometinib (VS-6766) monotherapy or avutometinib (VS-6766) in combination with defactinib, in KRAS-G12V NSCLC | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1
To evaluate the initial efficacy of avutometinib (VS-6766) in combination with defactinib in BRAF-MT NSCLC | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1
To determine efficacy in KRAS-other (non-G12V) NSCLC | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1
To determine the efficacy of avutometinib (VS-6766) in combination with defactinib in BRAF-MT NSCLC | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1

SECONDARY OUTCOMES:
To characterize the safety and toxicity profile of VS-6766 as a monotherapy and in combination with defactinib in KRAS-MT NSCLC and in BRAF-MT NSCLC | 24 weeks
  Adverse events (AEs), serious AEs (SAEs), vital signs, physical examinations, clinical laboratory values, and tolerability (dose interruptions/reductions)
Overall Response Rate per RECIST 1.1 as assessed by Investigator | From start of treatment to confirmation of response; 24 weeks
  Proportioned subjects achieving a CR or PR as assess by the investigator
Duration of Response (DOR) | Time from the first documentation of response to first documentation of progressive disease or death due to any cause, greater than or equal to 6 months
  Time of first response to PD as assessed by the IRC
Disease Control Rate (DCR) | Greater than or equal to 8 weeks
  CR and PR stable disease as assessed by the IRC
Progression Free Survival (PFS) | Up to 5 years
  From the time of first dose of study intervention to PD or death from any cause
Overall Survival (OS) | Up to 5 years
  From time of first dose of study intervention to death

CONTACTS AND LOCATIONS:
Overall Officials: Ross Camidge, MD, PhD, Principal Investigator — University of Colorado, Denver; MD Verastem, Study Director — Verastem, Inc.
Locations (45):
- United States (28):
  - City of Hope, Duarte, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center-Duchossois Center for Advanced Medicine, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Hematology/Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Maryland Oncology Hematology P.A, Columbia, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute/Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health-Monter Cancer Center, Lake Success, New York
  - Zangmeister Cancer Center, Columbus, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Univ. of Pittsburgh Med Center, Pittsburgh, Pennsylvania
  - Chattanooga Oncology Hematology Assoc., Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Texas Oncology Ft Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology, Grapevine, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- France (5):
  - Centre Leon Berard, Lyon
  - Hopital Nord Marseille, Marseille
  - Hopital Cochin, Paris
  - Institute De Cancerologie De L'Ouest Site Paul Papin Oncologie Medicale, Saint-Herblain
  - Cancerologie Gustave Roussy - Cancer Medicine, Villejuif
- Germany (3):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinkum Leipzig, Leipzig
  - Evangelisches Klinkum Bethel, Straße
- Italy (4):
  - Azienda Ospedaliera Universitaria, Orbassano, Torino
  - Irccs, Irts, Meldola
  - UOC di Oncologia Medica, Parma
  - Centro Ricerche Cliniche di Verona, Verona
- Spain (5):
  - Complejo Hospitalario Universiario a Coruna Teresa, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital 12 de Octubre, Córdoba
  - Universitario de Teatinos, Málaga
  - Hospital Universitario Virgen de la Macarena, Seville

REFERENCES:
- [Derived] Capelletto E, Bironzo P, Denis L, Koustenis A, Bungaro M, Novello S. Single agent VS-6766 or VS-6766 plus defactinib in KRAS-mutant non-small-cell lung cancer: the RAMP-202 phase II trial. Future Oncol. 2022 May;18(16):1907-1915. doi: 10.2217/fon-2021-1582. Epub 2022 Mar 14. PMID 35285277